CLINICAL TRIAL: NCT01120951
Title: Clinical Assessment of the Use of the R8 Respiratory Rate Counter in Post-Operative Recovery in Adults and Adolescents
Status: Completed | Type: Observational
Sponsor: Anaxsys Technology Ltd (Industry)
Responsible Party: Dr Ian Smith, Directorate of Anaesthesia, University Hospital of North Staffordshire, UK
Other Study IDs: ATL01009
Record Dates: First submitted 2010-05-09; First posted 2010-05-11 (Estimated); Last update posted 2010-05-18 (Estimated); Status verified 2010-05

CONDITIONS: Respiratory Rate Changes
Keywords: Respiratory rate R8 Anaxsys

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The study aims to to establish whether or not measurement of respiratory rate taken using the Anaxsys Technology Ltd Respiratory Counter (R8 Counter) are equivalent to manual respiratory rate counting methods in patients receiving oxygen via a face mask.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged 12 years and above following elective surgery under general anaesthesia

Exclusion Criteria:

* Patients admitted for emergency surgery
* Patients having ASA rating of 3 or greater
* Patients not receiving general anaesthesia
* Patients expected to be in post-operative recovery for less than 15 minutes

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Male or female patients aged 12 years and above following elective surgery under general anaesthesia
Sampling Method: Non-Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2010-01; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United Kingdom (4):
  - Papworth Hospital NHS Foundation Trust, Cambridge, Cambridgeshire
  - University Hospital of North Staffordshire, Stoke-on-Trent, Staffordshire
  - St. Peter's and Ashford Hospital NHS Trust, Guildford, Surrey
  - Russells Hall Hospital, Dudley, West Midlands